CLINICAL TRIAL: NCT03518294
Title: NASH Fitness Intervention in Thrombosis Trial (NASHFit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Stine, Assistant Professor Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8507
Record Dates: First submitted 2018-04-23; First posted 2018-05-08 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Liver Diseases; Blood Disorder; Digestive System Disease
Keywords: NAFLD; NASH
MeSH Terms: conditions — Liver Diseases; Hematologic Diseases; Digestive System Diseases; Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Standard of care Aerobic exercise
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Subjects in the control condition will be instructed to continue their medical care at the discretion of their treating medical professional. They will be informed to maintain their current physical activity level. Weekly phone calls will be performed by study personnel to ensure adherence to the protocol (no changes in activity). Subjects will report to Penn State on a monthly basis for anthropometric assessment to confirm their self-reports and study investigators will perform and interim history and physical examination at that time.
- Aerobic Exercise (Experimental): Subjects in the aerobic exercise group will be supervised to exercise 30 minutes, 5 times per week at a moderate intensity. Formal exercise instruction and supervision will be provided by ACSM certified fitness professionals at the Penn State University Fitness Center. Aerobic exercise can be completed on either the treadmill, exercise bike, rowing machine or the elliptical machine.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Subjects in the aerobic exercise group will be supervised to exercise 30 minutes, 5 times per week at a moderate intensity. Formal exercise instruction and supervision will be provided by ACSM certified fitness professionals at the Penn State University Fitness Center. Aerobic exercise can be completed on either the treadmill, exercise bike, rowing machine or the elliptical machine.
  Arms: Aerobic Exercise

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the leading cause of chronic liver disease in the United States. The most advanced forms of NAFLD are associated with increased liver-related mortality and lower overall survival. The current standard of care for NAFLD is lifestyle changes through diet and exercise. The human genome and regulation of gene expression is influenced by physical activity. NAFLD is a prothrombotic state with derangements in all three phases of hemostasis leading to clinically important clotting events. Exercise can improve coagulation in healthy persons. In this proposal, we seek to begin a line of work to answer the question "Can lifestyle changes effectively mitigate the increased risk of clotting in patients with NAFLD?" focusing initially on the at-risk population genetically susceptible to advanced disease.

DETAILED DESCRIPTION:
Often comorbid with obesity, nonalcoholic fatty liver disease (NAFLD) is the leading cause of chronic liver disease in the United States affecting 75-100 million adults, of which 15-20 million have the more severe variant nonalcoholic steatohepatitis (NASH). Conservative estimates project a doubling in NASH by 2025.The most advanced forms of NAFLD are associated with increased liver-related mortality and lower overall survival. The most effective treatment for NAFLD remains adopting healthy dietary and exercise patterns, however NAFLD patients are among the least physically active individuals. Predicting exercise behavior on an individual level is highly complex due to differing motivation, physiologic response to and subjective experience of exercise as well as emerging genetic evidence. The human genome and regulation of gene expression is influenced by physical activity. Patatin like phospholipase-3 (PNPLA3) rs738409 polymorphism (GG, GC and CC genotypes) plays a crucial role in the development of NAFLD. The GG genotype is both associated with advanced NAFLD, and predicts response to physical activity. Patients with NASH have extensive extrahepatic disease and are hypercoagulable. NASH is a prothrombotic state with fibrinolytic dysfunction through elevated plasminogen activator inhibitor (PAI-1), an independent risk factor for venous thromboembolism (VTE). Consequently, patients with NASH are predisposed to VTE; the risk of portal vein thrombosis (PVT) in NASH is 210% greater than in other liver disease. NASH patients are also at increased risk for pulmonary embolism (PE) and deep vein thrombosis (DVT).The most advanced forms of NASH have the greatest thrombotic risk. While studies observe that change in diet, weight and physical activity patterns improve NASH, it is not clear whether these lifestyle changes also reduce the elevated clot risk, however, moderate-intensity exercise leads to improved fibrinolysis in healthy persons.The NASHFit study is being done to find out if exercise is beneficial in decreasing the risk of clotting problems in patients with NASH. Exercise has been shown to decrease markers of clotting in healthy individuals as well as in those with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria Adults age >=18 or <70 years Liver biopsy <= 6months prior to enrollment Biopsy proven NASH(79)

Lack of secondary causes of hepatic fat accumulation:

Significant alcohol consumption (<21 drinks/week for men and <14 drinks/week for women) Chronic hepatitis C Wilson disease Lipodystrophy Parenteral nutrition Long-term use of steatogenic medications (mipomersen, lomitapide, amiodarone, methotrexate, tamoxifen, corticosteroids) Monogenic hereditary disorders

Exclusion Criteria >90 minutes/week of at least moderate intensity exercise over the previous three months Pregnancy BMI <18 or >40 kg/m2(16) Uncontrolled diabetes (changes in medication dosing over the previous three months or hemoglobin A1c >9%)(12) Active cardiac symptoms Severe medical comorbidities/psychiatric illness Decompensated cirrhosis (history of esophageal varices, ascites or hepatic encephalopathy) Abdominal hernia Cancer with life expectancy <6 months MRI contraindications (severe claustrophobia, implanted ferrous metal) Other liver disease (positive hepatitis B surface antigen, antinuclear antibody titer >1:160) Active weight-loss program participation or weight-loss supplement use Active substance abuse/smoking Inability to provide informed consent Institutionalized/prisoner Inability to walk > 2 blocks or ¼ mile. Physical Activity Readiness Questionnaire (PAR-Q) score >=1 at the discretion of the study PI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Stine, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Channapragada T, Batra S, Hummer BL, Chinchilli VM, Huang D, Loomba R, Schreibman IR, Stine JG. Aerobic Exercise Training Leads to MASH Resolution as Defined by the MASH Resolution Index. Dig Dis Sci. 2025 Sep 3. doi: 10.1007/s10620-025-09361-9. Online ahead of print. PMID 40900364
- [Derived] Motz V, Faust A, Dahmus J, Stern B, Soriano C, Stine JG. Utilization of a Directly Supervised Telehealth-Based Exercise Training Program in Patients With Nonalcoholic Steatohepatitis: Feasibility Study. JMIR Form Res. 2021 Aug 17;5(8):e30239. doi: 10.2196/30239. PMID 34402795

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 patients were screened for this study. Three were excluded after screening (two declined and one was excluded because they were actively smoking)
Period: Overall Study
Arm/Group | Standard of Care | Aerobic Exercise
Started | 10 | 18
Completed | 8 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Aerobic Exercise | Total
Number analyzed (Participants) | 10 | 18 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 18 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 12 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 17 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 18 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 18 | 28

OUTCOME MEASURES:

1. Primary Outcome: PAI-1 Level
Description: Change in fibrinolysis as indicated by PAI-1 level was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 8 | 16
ng/mL | 151.4 (51.5) | 176.2 (71.9)

2. Secondary Outcome: Change in Von Williebrand Factor (vWF)
Description: Change in vWF was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: International Units/Liter
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
International Units/Liter | 140.1 (63.1) | 128.4 (39.8)

3. Secondary Outcome: Change in Protein S
Description: Change in protein S was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
IU/dL | 106.3 (24.6) | 101.5 (22.4)

4. Secondary Outcome: Change in Factor VIII
Description: Change in factor VIII was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: International Units/Liter
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
International Units/Liter | 210.0 (75.0) | 188.6 (66.4)

5. Secondary Outcome: Change in Fibrinogen
Description: Change in fibrinogen was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
mg/dL | 352.4 (56.1) | 377.2 (83.5)

6. Secondary Outcome: Change in Antithrombin
Description: Change in antithrombin was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: percentage of protein
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
percentage of protein | 95.6 (12.1) | 102.2 (15.6)

7. Secondary Outcome: Change in Protein C
Description: Change in protein C was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
IU/dL | 169.0 (50.6) | 152.6 (55.9)

8. Secondary Outcome: Change in Adiponectin
Description: Change in adipontin was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
ng/mL | 3482.3 (1728.8) | 1065.1 (1220.7)

9. Secondary Outcome: Patatin Like Phospholipase-3 (PNPLA3) rs738409 Polymorphism
Description: Patatin like phospholipase-3 (PNPLA3) rs738409 polymorphism genotyping subjects (GG, GC and CC genotypes)
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
Participants
  CC | 3 | 8
  GC | 5 | 5
  GG | 2 | 5

10. Secondary Outcome: Change in PAI-1 Stratified by Fibrosis Stage
Description: Change is the difference between measurements at baseline and 5 months
Time Frame: 5 months
Population: The intended analysis was not performed for both groups, and instead this subset analyzed exercise group participants only.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- F0/F1; F2 Fibrosis; F3 Fibrosis: fibrosis stage
Arm/Group | F0/F1 | F2 Fibrosis | F3 Fibrosis
Number analyzed (Participants) | 12 | 2 | 4
ng/mL
  Baseline | 176.7 (120.9) | 241.4 (4.8) | 131.7 (24.4)
  Post exercise | 122.7 (36.6) | 196.1 (46.5) | 127.8 (36.7)

11. Secondary Outcome: Change in % Hepatic Fat
Description: Change in % hepatic fat was calculated by taking the difference of measurements at baseline and 5 months.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: percentage of liver
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
percentage of liver | 22.5 (10.5) | 20.4 (7.7)

12. Secondary Outcome: Health Related Quality of Life (HRQOL) Change
Description: Data was collected at baseline and at 5 months to assess changes in domains of health.
  PROMIS-29 Profile v2.1 (Physical function & pain interference) PROMIS Bank v2.0 - Instrumental Support (Social Support)
  Scores are reported as standardized T-score metrics derived from population means, with a mean of 50 and standard deviation of 10. The minimum is 0 and the maximum is 90.
  A higher score for fatigue, pain intensity, pain interference, sleep disturbance, anxiety and depression means a worse outcome.
  A higher score for physical function and social roles means a better outcome.
Time Frame: 5 months (20 weeks)
Population: ITT
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Standard of Care | Aerobic Exercise
Number analyzed (Participants) | 10 | 18
T-score
  Physical function | -2.5 (6.5) | 1.5 (5.0)
  Pain interference | 4.3 (9.6) | -3.4 (5.6)
  Social support | -0.7 (6.6) | 5.0 (7.0)

ADVERSE EVENTS:
Time Frame: up to 5 months
Arm/Group | Standard of Care | Aerobic Exercise
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/18
Other Adverse Events (participants affected / at risk) | 1/10 | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=10) | Aerobic Exercise (N=18)
Partial Knee Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) — A standard of care control subject elected to have knee surgery to treat longstanding osteoarthritis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=10) | Aerobic Exercise (N=18)
AEs (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)

LIMITATIONS AND CAVEATS:
Possible limitations include the sample size, lack of allocation concealment, study population largely of early-stage NASH that was also predominantly non-Hispanic white, lack of histologic endpoint, lack of long-term clinical outcomes and inability to show global changes in hemostasis with TEG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT03518294/Prot_SAP_000.pdf